CLINICAL TRIAL: NCT05513768
Title: Can First Trimester Serum Myocine Binding Protein c Level Predict Preterm Birth
Brief Title: PRETERM DELİVERY and MYOCINE BINDING PROTEIN C LEVELs
Status: Completed | Type: Observational
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, Elif Yıldız, MEDİCAL DOCTOR, Gaziosmanpasa Research and Education Hospital
Other Study IDs: GaziosmanpasaTREHKHD
Record Dates: First submitted 2022-08-22; First posted 2022-08-24 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Preterm
Keywords: PRETERM DELİVERY, MBPC,
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- women who gave birth prematurely: women who had serum taken in the first trimester and gave birth earlier than 37 weeks according to the time of delivery
  Interventions: Diagnostic Test: level of myosin binding protein c in serum
- those who gave birth on time: women who have had serum taken in the first trimester, stored and delivered on time
  Interventions: Diagnostic Test: level of myosin binding protein c in serum

INTERVENTIONS:
Diagnostic Test: level of myosin binding protein c in serum — Serum samples will be taken from the participants in the first trimester, transferred to eppendorf tubes after appropriate procedures, and stored at -80 degrees until the time of deliveryParticipants will be divided into two groups according to the timing of birthThe first group is those who gave birth earlier than 37 weeks those who gave birth on time in the other group The mbpc levels will be looked at and compared.

SUMMARY:
IT WAS AIMED TO EVALUATE IF MBPC CAN BE USED IN PREDICTION OF EARLY BIRTH. TAKING THE FIRST TRIMESTER FROM PREGNANCY WAS STORED UNTIL THE TIMING OF DELIVERY.THE PARTICIPANTS WERE SEPARATED INTO TWO GROUPS ACCORDING TO THE TIME OF BIRTH, EARLY AND TIMELY.

SERUM MBPC LEVELS BETWEEN TWO GROUPS EVALUATED.

DETAILED DESCRIPTION:
IT WAS AIMED TO EVALUATE IF MBPC CAN BE USED IN PREDICTION OF EARLY BIRTH. TAKING THE FIRST TRIMESTER FROM PREGNANCY WAS STORED UNTIL THE TIMING OF DELIVERY.THE PARTICIPANTS WERE SEPARATED INTO TWO GROUPS ACCORDING TO THE TIME OF BIRTH, EARLY AND TIMELY.

SERUM MBPC LEVELS BETWEEN TWO GROUPS EVALUATED.A TOTAL OF 90 WOMEN WERE PLANNED TO INCLUDE 45 STUDY 45 CONTROL GROUP IN THE STUDY.

ELIGIBILITY:
Inclusion Criteria:

* being pregnant in the first trimester
* be between 18-40 years old

Exclusion Criteria:

* no history of preterm birth
* being pregnant with assisted reproductive techniques
* having a multiple pregnancy
* have cervical insufficiency

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Includes participants whose serum samples were collected in the first trimester, stored, and then divided into two according to timing of delivery fırst grup ıs preterm group, and second one ıs those who gave birth on time
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
detection of prediction value of serum mbpc levels in preterm delivery | 10 mounths
  identifying prediction value of first trmester serum mbpc levels by comparing by serum levels of mbpc in groups

CONTACTS AND LOCATIONS:
Overall Officials: elif yıldız, Principal Investigator — Gaziosmanpasa Research and Education Hospital
Locations (1):
- Gaziosmanpasa Training and Research Hospital, Istanbul, Gaziosmanpaşa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No